CLINICAL TRIAL: NCT06052501
Title: 3D Evaluation of the Lip Support in a Full-arch Implant-supported Rehabilitations
Status: Recruiting | Type: Observational
Sponsor: Implantology Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DMarques
Record Dates: First submitted 2023-09-19; First posted 2023-09-25 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Digital Technology; Prosthesis User; Lip; Oral Soft Tissue Conditions; Occlusion
Keywords: three-dimensional imaging; prosthodontics; full-arch; facial scanner
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia; Bites and Stings

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Removable of the full arch implant-supported prostheses — The intervention planned will be the removal of full arch implant-supported prostheses and the acquisition of a digital image through a facial scanner before and after this moment.

SUMMARY:
The goal of this observational study is to evaluate the impact of a full arch implant-supported prostheses in the lip support. In a complex rehabilitation cases, the process between the diagnosis and the delivery of a prostheses may lead with many clinical and laboratorial choices which influence the final design of the prosthetic work and consequently the facial profile of the patient.

The use of 3D facial scanners and advanced superimposition methodology allows the investigators to objectively measure several relevant parameters such as vertical occlusion of dimension and lip support.

DETAILED DESCRIPTION:
Digital technologies have evolved exponentially in the dental medicine field endorsing a change between the conventional methods to virtually based methodologies in daily clinical and laboratorial practice.

Combining facial aspects and proportions with dento-gingival parameters are the basis when planning a new smile design and a final rehabilitationFacial surface images can be used for more predictable measurement and quantification of vertical dimension of occlusion and lip support before, during and after a full mouth rehabilitation. Besides that, the information obtained by facial scanners have a major impact in treatment planning process especially in multidisciplinary complex cases with the simulation of the treatment, identification of patient's expectations and the implementation of an effective communication tool.

The 4D-virtual patient is the future regarding the management of a patient in dental medicine, since the beginning of the process with data acquisition for the diagnosis to the definitive oral rehabilitation procedures. Similar to any methodology, it is important to understand what are the basis of the facial scanning and what protocols can obtain better results in terms of accuracy and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with at least a full-arch implant supported rehabilitation in the upper arch
* Individuals with a provisional or a definitive implant-supported prosthesis
* Individuals with a stable occlusion function
* Individuals with compliance to collaborate with the research protocol

Exclusion Criteria:

* Individuals with history of hypersensitivity to external light or any similar condition
* Individuals in an active surgical treatment period
* Individuals in an active orthodontic treatment in the opposite arch
* Individuals in an active facial treatment
* Individuals who did not attend the maintenance visits

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients from private clinic in which the implant treatment was performed. These patients must have their maintenance appointments up to date.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Volumetric changes in peri-oral area | same day
  The primary outcome is to evaluate the changes in volume in peri-oral area after removal a full arch implant-supported prostheses according to a digital analysis (RMS)

SECONDARY OUTCOMES:
Distance between the upper lip and E-line in sagital profile | same day
  The secondary outcome is to quantify the changes in the distance between the upper lip and the Rickett's Aesthetic Line (E-line)
Distance between the lower lip and E-line in sagital profile | same day
  The third outcome is to quantify the changes in the distance between the lower lip and the Rickett's Aesthetic Line (E-line)
Naso-labial angle | same day
  The fourth outcome is to quantify the changes in the naso-labial angle related to the absence of the fixed prostheses

OTHER OUTCOMES:
Confounding factors | same day
  Type of definitive rehabilitation, time of implant surgery, extension of rehabilitation/edentulism

CONTACTS AND LOCATIONS:
Overall Officials: João Caramês, DDS, PhD, Study Director — Implantology Institute; Duarte Marques, DDS, PhD, Study Chair — Implantology Institute; Rita Alves, DDS, Principal Investigator — Implantology Institute
Locations (1):
- Implantology Institute, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No